CLINICAL TRIAL: NCT03286920
Title: Effect of Postoperative Family Nutrition Mode on Weight/BMI of Patients With Esophageal Cancer
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Cancer Hospital & Institute (Other)
Collaborators: Sun Yat-sen University (Other); Zhejiang Cancer Hospital (Other); Shanghai Chest Hospital (Other); China-Japan Friendship Hospital (Other); Fudan University (Other); Shandong Provincial Hospital (Other Government); Hebei Medical University Fourth Hospital (Other); Anyang Tumor Hospital (Other); The First Affiliated Hospital of Anhui Medical University (Other); The First Affiliated Hospital of Bengbu Medical University (Other); Tongji Hospital (Other); Shanxi Province Cancer Hospital (Other); The Third Affiliated Hospital of Harbin Medical University (Other); Liaoning Cancer Hospital & Institute (Other); Wuhan General Hospital of Guangzhou Military Command (Other); Second Xiangya Hospital of Central South University (Other); The First Hospital of Jilin University (Other); Chinese PLA General Hospital (Other); Hunan Provincial People's Hospital (Other); Fujian Cancer Hospital (Other Government); Qilu Hospital of Shandong University (Other); Union hospital of Fujian Medical University (Other); Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Principal Investigator, Ke-Neng Chen, MD, PhD, FRCS, Doctor, Peking University Cancer Hospital & Institute
Other Study IDs: 2017-06-01
Record Dates: First submitted 2017-09-15; First posted 2017-09-19 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Esophageal Cancer
Keywords: home nutrition; BMI; postoperative; body weight
MeSH Terms: conditions — Esophageal Neoplasms; Body Weight

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Oral natural diet: As for patients in oral natural diet group, the the participants shall receive oral natural diet.
- Oral nutrition supplement group: As for patients in oral nutrition supplement group, in addition to oral natural die, the participants shall receive oral enteral supplement providing 750-1500kcal/d.
  Interventions: Dietary Supplement: Oral nutrition supplement
- Tube feeding nutrition supplement group: As for patients in tube feeding group, in addition to oral natural die, the participants shall receive tube feeding nutrition supplement providing 750-1500kcal/d.
  Interventions: Dietary Supplement: Tube feeding nutrition supplement

INTERVENTIONS:
Dietary Supplement: Oral nutrition supplement — As for patients in oral nutrition supplement group, in addition to oral natural die, the participants shall receive oral enteral supplement providing 750-1500kcal/d.
  Groups: Oral nutrition supplement group
Dietary Supplement: Tube feeding nutrition supplement — As for patients in tube feeding group, in addition to oral natural die, the participants shall receive Tube feeding nutrition supplement providing 750-1500kcal/d.
  Groups: Tube feeding nutrition supplement group

SUMMARY:
This clinical trial is designed to be a multi-center prospective observational study which shall compare the effect of different postoperative home nutrition modes on recent nutritional index (weight/BMI) of patients with esophageal cancer and recent outcomes. Different postoperative home nutrition modes adopted in this study includes oral natural diet, oral nutrition supplement and tube feeding.

DETAILED DESCRIPTION:
STUDY BACKGROUND Esophageal cancer is a common cancer in China and due to its influence on diet intake, patients with esophageal cancer are often combined with nutrition deficiency, which causes relatively high nutrition risk to treatment. Studies conducted by Martin et al showed that the degree of body weight loss in patients with malignancy is related to BMI level and prognosis. The patients with severe body weight loss and low BMI have poor prognosis, especially for patients with esophageal cancer.

At present, perioperative nutrition support for patients with esophageal cancer has been recognized and has been recommended as routine in 2017 NCCN guideline. How to implement good home nutrition within one month after patient discharge and recover nutrition index as soon as possible has become a focus for esophageal surgeon.

Many clinical trials have already investigated enteral nutrition support approach during anti-cancer treatment period in patients with malignancy. However, only a few clinical trials are good designed. Therefore the investigators hope to via this multi-center prospective observational study to provide evidence for this question.

OBJECTIVES:

1. To explore the relationship between postoperative home nutrition support treatment approach and nutritional status of patients with esophageal cancer;
2. To explore the relationship between postoperative home nutrition support treatment approach and recent prognosis in patients with esophageal cancer;
3. To promote the standardized application of postoperative home nutrition support treatment for patients with esophageal cancer.\

OUTLINE:

Included patients shall be divided into three groups according to the treatment plan of all centers, including oral natural diet, oral nutrition supplement and tube feeding. As for patients in oral natural diet group, the patients shall receive oral natural diet. As for patients in oral nutrition supplement group, in addition to oral natural die, the participants shall receive oral enteral supplement providing 750-1500kcal/d. As for patients in tube feeding group, in addition to oral natural die, the participants shall receive tube feeding enteral supplement providing 750-1500kcal/d.

All the included patients shall be followed up weekly within 1-3 weeks after discharge via telephone, at Day 30 after discharge and at Day 90 after discharge to assess the effectiveness and safety of different home nutrition supplement approaches.

PROJECTED ACCRUAL: A total of 600 patients will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

* Age below 80 years old;
* Esophageal cancer;
* Radical surgery;
* Normal gastrointestinal function

Exclusion Criteria:

* Patients with diabetes and poor blood glucose control;
* Patients with severe postoperative complications;
* Patients who can't tolerate lactose;
* Patients who decline inclusion and follow-ups

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with esophageal cancer who undergo surgery
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2017-09-20 (Actual); Primary Completion 2018-09 (Estimated); Study Completion 2018-09 (Estimated)

PRIMARY OUTCOMES:
Percentage of 5% body weight loss on Day 30 | Day 30 after discharge
  Percentage of 5% body weight loss on Day 30 compared to the body weight at discharge

SECONDARY OUTCOMES:
Completion ratio of different nutrition support approaches | Day 30 after discharge
  Completion ratio of different nutrition support approaches
Quality of life assessment using EORTC QLQ-C30 scale and QLQ-OG25 scale | Day30 and Day 90
  Assessment on patients' quality of life using EORTC QLQ-C30 scale and QLQ-OG25 scale in different nutrition support approach groups and investigate the relationship between different nutrition support approaches and patients' quality of life
Complications of home enteral nutrition support | Day30
  Assessment on complications of home enteral nutrition support
Delay and interruption ratio of adjuvant treatment | Day 30 and Day 90
  Delay and interruption ratio of adjuvant treatment including whether chemotherapy and radiotherapy can be implemented on time
Re-hospitalization ratio | Day 90
  Re-hospitalization ratio within 90 days after discharge

CONTACTS AND LOCATIONS:
Overall Officials: Keneng Chen, M.D., Principal Investigator — Peking University Cancer Hospital & Institute
Locations (23):
- China (23):
  - First Affiliated Hospital Bengbu Medical College, Bengbu, Anhui
  - The First Affiliated Hospital of Anhui Medical University, Hefei, Anhui
  - Beijing Cancer Hospital, Beijing, Beijing Municipality
  - China-Japan Friendship Hospital, Beijing, Beijing Municipality
  - Chinese PLA General Hospital, Beijing, Beijing Municipality
  - Daping Hospital and the Research Institute of Surgery of the Third Military Medical University, Chongqing, Chongqing Municipality
  - Union hospital of Fujian Medical University, Fuzhou, Fujian
  - Sun Yat-sen University Cancer Hospital, Guangdong, Guangdong
  - Guangzhou General Hospital of Guangzhou Military Command, Guangzhou, Guangdong
  - Hebei Medical University Fourth Hospital, Shijiazhuang, Hebei
  - The Third Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Anyang Tumor Hospital, Anyang, Henan
  - Tongji Hospital, Wuhan, Hubei
  - Second Xiangya Hospital of Central South University, Changsha, Hunan
  - First Hospital of Jilin University, Changchun, Jilin
  - Liaoning Tumor Hospital & Institute, Shenyang, Liaoning
  - Qilu Hospital of Shandong University, Jinan, Shandong
  - Shandong Provincial Hospital, Jinan, Shandong
  - Fudan University Cancer Hospital, Shanghai, Shanghai Municipality
  - Shanghai Chest Hospital, Shanghai, Shanghai Municipality
  - Shanxi Province Cancer Hospital, Taiyuan, Shanxi
  - First People's Hospital of Yunan province, Kunming, Yunan
  - Zhejiang Cancer Hospital, Hanzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: No